CLINICAL TRIAL: NCT04002453
Title: Outpatient Parenteral Antibiotic Therapy in the Metropolitan Area of Cologne
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Clara Lehmann, Head of outpatient clinic, University of Cologne
Other Study IDs: C-OPAT
Record Dates: First submitted 2019-06-21; First posted 2019-06-28 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Implementation of OPAT in Germany
Keywords: OPAT; infectious diseases; implementation
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatient parenteral antimicrobial therapy: Patients with an infectious disease that receive an outpatient parenteral antimicrobial therapy
  Interventions: Procedure: Outpatient Parenteral Antibiotic Therapy

INTERVENTIONS:
Procedure: Outpatient Parenteral Antibiotic Therapy — Application of outpatient parenteral antibiotic therapy in patients with infectious diseases to allow them to get discharged from hospital.

SUMMARY:
Many infectious diseases require a therapy that is administered intravenously due to a lack of oral treatments. Affected patients often have to stay weeks or even months in hospital just for receiving their therapy although they do not feel severely unwell.

Outpatient parenteral antibiotic therapy (OPAT) allows these patients under certain requirements to get discharged from hospital and apply the antibiotic treatment on their own. For these patients quality of life improves by feeling more comfortable at home and being able to participate in everyday life or even go back to work. For the hospitals a reduced inpatient health care means a clear reduction of costs.

The benefits of OPAT are obvious, shown by several studies, and in many countries e.g. the USA OPAT is a very well established way of treatment. In Germany however OPAT is used very infrequently and not in a standardized manner. This is probably due to inadequate knowledge of this form of treatment and deficits in the outpatient care structure, as OPAT is not reflected in the remuneration system of the German health care system despite internationally proven benefits.

The aim of this study is to identify and analyze possible obstacles to the implementation of OPAT into the standard patient care in Germany regarding financial, structural and medical limitations. Therefore the investigators intend to treat 120 patients in the metropolitan area of Cologne with OPAT and observe effectiveness, safety, logistics and acceptance to this kind of therapy.

If successful, the project should help to identify the potential of OPAT for Germany. If positive effects and feasibility can be demonstrated in the Cologne metropolitan region, OPAT could become an important therapy option with many advantages for certain patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who get OPAT

Exclusion Criteria:

* patients who don't get OPAT or are not capable to give their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic, university hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with effective OPAT | 12 weeks
  Successful administration and completion of the antiinfective therapy
Number of Patients With Treatment-Related Adverse Events | 12 weeks
  side-effetcs of treatment and catheter-related infections

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peter S, Oberrohrmann C, Pfaff H, Lehmann C, Schmidt-Hellerau K, Brandes V, Leisse C, Lindemann CH, Ihle P, Kupper-Nybelen J, Hagemeier A, Scholten N. Exploring patients' perspectives: a mixed methods study on Outpatient Parenteral Antimicrobial Therapy (OPAT) experiences. BMC Health Serv Res. 2024 Apr 29;24(1):544. doi: 10.1186/s12913-024-11017-9. PMID 38685017
- [Derived] Schmidt-Hellerau K, Baade N, Gunther M, Scholten N, Lindemann CH, Leisse C, Oberrohrmann C, Peter S, Jung N, Suarez I, Horn C, Ihle P, Kupper-Nybelen J, Hagemeier A, Hellmich M, Lehmann C. Outpatient parenteral antimicrobial therapy (OPAT) in Germany: insights and clinical outcomes from the K-APAT cohort study. Infection. 2024 Aug;52(4):1407-1414. doi: 10.1007/s15010-024-02199-9. Epub 2024 Mar 13. PMID 38478255
- [Derived] Scholten N, Leisse C, Brandes V, Oberrohrmann C, Ihle P, Peter S, Hagemeier A, Hellmich M, Lindemann CH, Samel C, Pfaff H, Lehmann C. Outpatient parenteral antimicrobial therapy in Germany: a prospective cohort study protocol. BMJ Open. 2022 Nov 14;12(11):e061417. doi: 10.1136/bmjopen-2022-061417. PMID 36375971